CLINICAL TRIAL: NCT05398250
Title: A Comparison of Two Brief Suicide Prevention Interventions Tailored for Youth on the Autism Spectrum
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Pennsylvania (Other); Nationwide Children's Hospital (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Children's Hospital of Philadelphia (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-2110
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Suicidal Ideation; Suicidal and Self-injurious Behavior; Suicide; Autism Spectrum Disorder
Keywords: Suicide Prevention; Autism Spectrum Disorder; Safety Planning Intervention
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior; Suicide; Autism Spectrum Disorder; Suicide Prevention | interventions — lambda Spi-1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning Intervention Tailored for Autistic Individuals (Active Comparator): The Safety Planning Intervention Tailored for Autistic individuals (SPI-A) is a brief collaborative intervention that results in an individually tailored plan designed to lower the short-term risk of suicide in autistic youth.
  Interventions: Behavioral: Safety Planning Intervention tailored for Autistic Individuals
- Safety Planning Intervention Tailored for Autistic Individuals Plus Structured Follow-Up Contacts (Active Comparator): The Safety Planning Intervention Tailored for Autistic individuals plus structured follow-up contacts (SPI-A+) is a multi-component intervention comprised of SPI-A and structured follow-up consisting of at least 2 brief contacts.
  Interventions: Behavioral: Safety Planning Intervention Tailored for Autistic Individuals Plus Structured Follow-Up Contacts

INTERVENTIONS:
Behavioral: Safety Planning Intervention tailored for Autistic Individuals — To develop the SPI-A, clinicians work collaboratively with patients, and when indicated, their family members, to create a list of concrete coping mechanisms to be enacted leading up to or during a crisis. This list can be depicted in writing or pictorially, depending on patient preference. As part of the intervention, patients (and family members, when appropriate) also identify warning signs that signal the need to use the safety plan, as well as a detailed plan for reducing access to lethal means. SPI-A is a stand-alone intervention without a follow-up component.
  Other Names: SPI-A
  Arms: Safety Planning Intervention Tailored for Autistic Individuals
Behavioral: Safety Planning Intervention Tailored for Autistic Individuals Plus Structured Follow-Up Contacts — SPI-A+ includes SPI-A plus a structured follow-up component. The structured follow-up component of SPI-A+ includes three elements:
  1. A brief risk assessment and mood check
  2. Review and, if needed, revision of SPI-A
  3. Support related to outpatient mental health treatment initiation
  Other Names: SPI-A+
  Arms: Safety Planning Intervention Tailored for Autistic Individuals Plus Structured Follow-Up Contacts

SUMMARY:
Rates of suicide have increased significantly over the past two decades, particularly among youth. Compared to the general population, autistic people are significantly more likely to think about suicide, attempt suicide, and die by suicide. Autistic individuals have identified suicide prevention as a top research priority; however, little is known about how to best help autistic youth at risk for suicide. The purpose of this study is to compare the effectiveness, feasibility, and acceptability of two suicide prevention strategies tailored for autistic individuals: the Safety Planning Intervention tailored for Autistic individuals (SPI-A) and SPI-A plus structured follow-up contacts (SPI-A+).

DETAILED DESCRIPTION:
**Participants**

Participants are from three distinct groups: health systems leaders, clinicians, and autistic youth (patients). The autistic youth participant pool is comprised of three subgroups, described below.

1. "Basic EHR-Only" Arm:

   Population: All individuals 12-24yo scheduled for a clinical visit with a consented clinician during the study recruitment period qualify for this arm. The total number of subjects for this subgroup is expected to exceed 15k individuals.

   Participation is limited to Electronic Health Record (EHR) review only. Participants will not have contact with the study team.
2. "Enhanced EHR-Only" Arm: Population: Individuals meeting the above criteria who also receive one of the interventions of interest (SPI-A or SPI-A+) during routine clinical care. Approximately 250-400 individuals are expected to qualify for this arm.

   Participation is limited to EHR review and abstraction to evaluate outcomes related to the SPI-A and SPI-A+ interventions. Participants will not have contact with the study team.
3. "Active Patient-Reported Outcomes (PRO)" Arm: Population: Individuals meeting the criteria for the "Enhanced EHR-Only" arm who are referred by a participating clinician to the study team and provide informed con/assent to participate in survey and interview data collection constitute this arm.

Participation consists of medical records review and abstraction, as well as survey and interview data collection. Please note that enrollment into this arm concluded 9/1/2025.

**Aims**

This study includes three aims:

Aim 1: Among autistic youth (age 12-24) at risk for suicide, compare the effectiveness of SPI-A vs. SPI-A+. The primary outcomes of interest are suicidal ideation (SI) and suicidal behavior (SB), as derived from electronic health records (EHR) and patient reported outcomes (PRO) data. Secondary patient-centered outcomes are mental health treatment initiation and engagement (EHR and PRO), use of acute care services for suicidality (EHR and PRO), quality of life (PRO), well-being (PRO), skills to manage SI (PRO), access to lethal means (PRO), and safety plan use (PRO).

Aim 2: Compare implementation outcomes of acceptability and feasibility for the two interventions from the perspectives of patients, clinicians, and health system administrators.

Aim 3: Explore patient characteristics that may moderate the relationship between intervention and SI and SB.

ELIGIBILITY:
(A) Patient Participants

Please note that that eligibility criteria differ for each distinct patient subgroup as defined below.

A.1 - Basic EHR-Only Arm

Inclusion criteria:

* 12-24 years old
* Scheduled for a clinical visit with a consented clinician Exclusion criteria: None

A.2 - Enhanced EHR-Only Arm:

Inclusion criteria:

* Meets inclusion criteria for the Basic EHR-Only arm
* Receives one of the interventions being studied (SPI-A or SPI-A+) as part of routine clinical care

Exclusion criteria: Presence of documentation that the patient declines all research participation

A.3 - Active PRO Arm:

Inclusion Criteria:

* Meets inclusion criteria for the Enhanced EHR-Only arm
* Referred to the study team by a consented clinician
* Able and willing to provide informed consent (age 18+) or assent and parental/guardian consent (age < 18)
* Able to speak English (and, if applicable, at least one guardian also able to speak English)

Exclusion Criteria: Altered mental status that precludes ability to provide informed assent or consent (acute psychosis, intoxication, or mania)

(B) Clinician Participants

Inclusion Criteria:

* Employment as a provider serving autistic patients at one of the study sites
* Employment in a role that involves suicide risk intervention with youth patients at a participating clinic
* Able to read and speak English
* Able and willing to provide informed consent

Exclusion Criteria: None

(C) Health System Leader Participants

Inclusion Criteria:

* Health system or clinic leader at one of the study sites
* Employed in a role that provides administrative oversight to clinicians conducting safety plans with patients
* Able to read and speak English
* Able and willing to provide informed consent

Exclusion Criteria: None

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1665 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation and behavior | Through 12 months of follow-up
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinical interview that measures suicidal ideation (range 0-5, with higher scores indicating more severe ideation) and suicidal behavior (count of total number of actual attempts, interrupted attempts, aborted attempts, and preparatory acts or behavior). The C-SSRS will be administered at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.

SECONDARY OUTCOMES:
Change in mental health treatment utilization | Up to 12 months
  The Service Assessment for Children and Adolescents (SACA) is an interview designed to gather information on the patient participants' use of mental health services, including residential (e.g., hospital), outpatient (e.g., outpatient mental health clinic), and school (e.g., counseling) services. The SACA will be administered at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Change in quality of life | Up to 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Autism Battery - Lifespan (PAB-L) is a subset of PROMIS measures that has been validated for assessment of quality of life among autistic individuals. The PAB-L youth self-report includes four domains: Subjective Well-being, Relationships, Emotional Distress, and Health. Items are rated on a 1-5 scale, with higher scores indicating a greater presence of the measured construct. Patient participants will complete the PAB-L at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Change in well-being | Up to 12 months
  Well-being will be measured with the Outcome Rating Scale (ORS), a 4-item visual analog scale assessing functioning in individual, interpersonal, social, and overall functioning over the past week. Item scores range from 0-10, with higher scores indicating better functioning. Patient participants will complete the ORS at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Change in skills to manage suicidal ideation | Up to 12 months
  The Suicide-Related Coping Scale (SRCS) assesses knowledge of and confidence in using coping strategies and supports to manage suicidal thoughts and urges. The SRCS items are rated on a 5-point scale ("strongly disagree" to "strongly agree"). Higher scores indicate greater coping skills to manage suicidal crises. Patient participants will complete the SRCS at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Change in access to lethal means | Up to 12 months
  The patient participants will answer the three access to lethal means questions from the Adapted Behavioral Risk Factor Surveillance System Survey (BRFSS), selected from the PhenX Toolkit, at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up. These questions capture whether firearms are present in the home and, if so, how they are stored (e.g., loaded and unlocked).
Change in safety plan use | Up to 12 months
  The Brief Safety Plan Use Scale (BSPUS) will be used to assess the extent to which patient participants have utilized their safety plans since the prior assessment timepoint (e.g., "How many times did you use the safety plan since last meeting?" "Where have you been keeping the safety plan?"). Patient participants will complete the BSPUS at 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Change in acute care services for suicidality | Up to 12 months
  The Service Assessment for Children and Adolescents (SACA) will be used to assess patient participants' acute care services for suicidal thoughts and behaviors. The SACA will be administered at baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up.
Intervention acceptability | Patient Participants: 1-month follow-up; Clinician and Health System Leader Participants: up to 4 years
  Patient, clinician, and health system leader participants will complete the Acceptability of Intervention Measure (AIM), a widely used four-item measure that can be administered to a wide range of stakeholders to determine the extent to which they believe an intervention is acceptable. Items are rated from 1-5, with higher scores indicating greater acceptability. Patient participants will complete the AIM at the 1-month follow-up timepoint. Clinician and health system leader participants will complete the AIM in Year 1 and Year 4 of the study.
Intervention feasibility | Patient Participants: 1-month follow-up; Clinician and Health System Leader Participants: up to 4 years
  Patient, clinician, and health system leader participants will complete the Feasibility of Intervention Measure (FIM), a widely used four-item measure that can be administered to a wide range of stakeholders to determine the extent to which they believe an intervention is feasible. Items are rated from 1-5, with higher scores indicating greater feasibility. Patient participants will complete the FIM at the 1-month follow-up timepoint. Clinician and health system leader participants will complete the FIM in Year 1 and Year 4 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Roubinov, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Shari Jager-Hyman, PhD, Principal Investigator — University of Pennsylvania
Locations (5):
- United States (5):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pennsylvania, Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that support the results will be shared after the publication of the final research report, for a period of at least 7 years, provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual data that support the results will be shared after the publication of the final research report, for a period of at least 7 years.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.